CLINICAL TRIAL: NCT05504733
Title: Evaluating the Functionality of a Novel Layperson Tourniquet: A Doppler Study
Brief Title: LAVA TQ Doppler Functionality Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: USUHS.2020-060; NM91959717 (Other Grant/Funding Number: Uniformed Services University of the Health Sciences)
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Traumatic Hemorrhage

STUDY DESIGN:
Intervention Model Description: This study will be a single blinded, randomized clinical trial.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Layperson Audiovisual Assist Tourniquet (LAVA TQ) (Experimental): For participants in the experimental arm, the Layperson Audiovisual Assist Tourniquet (LAVA TQ) is the first tourniquet applied to their leg as the intervention.
  Interventions: Device: Layperson Audiovisual Assist Tourniquet (LAVA TQ); Device: Combat Application Tourniquet
- Combat Application Tourniquet (CAT) (Active Comparator): For participants in the control/active comparator arm, the Combat Application Tourniquet (CAT) is the first tourniquet applied to their leg as the intervention.
  Interventions: Device: Layperson Audiovisual Assist Tourniquet (LAVA TQ); Device: Combat Application Tourniquet

INTERVENTIONS:
Device: Layperson Audiovisual Assist Tourniquet (LAVA TQ) — The Layperson Audiovisual Assist Tourniquet is a hemorrhage control device designed to occlude blood flow in the event of limb hemorrhage. This device provides audiovisual instructions and feedback.
Device: Combat Application Tourniquet — The Combat Application Tourniquet (CAT) is a hemorrhage control device designed to occlude blood blow in the event of a limb hemorrhage. The CAT utilizes a windlass rod design.

SUMMARY:
This is a single-blinded, randomized clinical trial to determine if the Layperson Audiovisual Assist tourniquet's (LAVA TQ) ability to occlude arterial blood flow is non-inferior to that of the Combat Application Tourniquet (CAT).

DETAILED DESCRIPTION:
1. Background and Significance

   Trauma is the leading cause of death in the United States for people ages 1 to 44; uncontrolled bleeding is a leading cause of those deaths.1 Immediate hemorrhage control, even prior to the arrival of emergency medical services, can save lives during these emergencies. Since the launch of the Stop the Bleed (STB) campaign in 2015, the public has been empowered to stop life-threatening hemorrhage.2 One of STB's five objectives is to equip every bleeding control kit with audio and visual instructions; this has not yet been achieved. Commonly used tourniquets, such as the Combat Application Tourniquet (CAT) or Special Operations Forces Tourniquet (SOF-T), do not provide audio instructions and are not designed to provide feedback to facilitate tourniquet application. A device that could facilitate application and provide real-time instructions and feedback could be immensely beneficial to both the public and the DoD, especially to minimally or untrained people such as DoD civilians, contractors, and dependents on military installations. To achieve the above mentioned STB's objective, the research team at the National Center for Disaster Medicine and Public Health is devoted to develop a layperson tourniquet with audio-visual instructions and performance feedback.

   In January 2020, the research team conducted a pilot study to evaluate this novel layperson tourniquet in a community lay public sample recruited from at the NBC Health Expo in Washington, DC. Findings of this pilot study were promising. One highlight of the results was that the proportion of participants who applied the tourniquet correctly using the layperson tourniquet was significantly higher than that using the CAT (93.3% versus 6.3%). Moreover, for when asked about their favoritism toward the tourniquet, 93.3% favored the novel layperson tourniquet, whereas 68.8% favored the CAT.

   In addition to research results, feedback provided by the participants in this pilot study allowed the research team and the manufacturing partner to make adjustments and improvements to the testing device. Now we have completed a pilot study evaluating overall user experience of the novel layperson tourniquet, our next step is to conduct a functionality study examining the function of this novel layperson tourniquet and to see if it performs on par with the CAT.
2. Objectives/Specific Aims/Research Questions

   The objective of the study is to determine if the Layperson Audiovisual Assist Tourniquet (LAVA TQ)'s ability to occlude arterial blood flow is non-inferior to a Combat Application Tourniquet (CAT).
3. Study Procedures

   This study will be a single blinded, randomized clinical trial. The study will be conducted in a room at USU's Multidisciplinary Laboratories.

   The study has two arms: SMART TQ is the experimental arm and CAT is the control arm. The study will consist of three groups of individuals:
   * Medical professionals who apply the tourniquet (we will call this group "medical professionals" in this protocol).
   * Volunteers who offer their legs for tourniquet application (we will call this group of individuals "study participants").
   * Blinded observers who will use a Doppler to check and monitor pulse. Absence of the dorsalis pedis pulse will be used to indicate occlusion of blood flow. The pulse monitored by the blinded observers will be used as an outcome for this research study. The only person blinded in the study will be the person checking for a successful application by measuring the doppler pulse - that is the blinded observers. There will be a bedsheet, or similar screen, placed between the portion of the participant's leg that has the tourniquet applied and the participant's foot where the doppler pulse will be measured. In addition, the research team will provide blinded observers noise-canceling headphones to minimize the influence of audio instructions provided by the LAVA TQ.

   We will recruit two medical professionals and two blinded observers and consent volunteers (i.e., participants).

   Two medical professionals will attend a training session prior to the study. The session will allow the study team to verify that medical professionals can apply both types of tourniquets successfully. We anticipate this training session lasting no more than one hour and will recruit one participant for the training session.

   Upon the completion of the informed consent, participants will be assigned study ID numbers. The study steps are below:
   * A study participant enters the study room, completing a demographic information sheet and taking blood pressure, and then lies down with the face and torso facing up.
   * To capture the baseline dorsalis pedis (DP) pulse: A blinded observer uses a doppler ultrasound to check DP pulse, the artery pulse on the surface of the foot. Doppler ultrasound is a small medical ultrasound machine that uses high-frequency sound waves to measure the amount of blood flow through the arteries and veins. The doppler ultrasound probe will be placed on the exposed foot, a pulse detected, and the location where the pulse is detected on that foot will be marked with an "X" using a surgical marker, and the doppler probed removed. This marked location will be where the doppler probe is placed later to determine whether there is a pulse.
   * The research team member will measure the circumference of the leg at the area of tourniquet application. To keep the application location consistent across all the participants, we will mark where on the leg the tourniquet should be placed for each application.
   * A medical professional records which leg will be used for tourniquet application (left leg or right leg).
   * The medical professional applies the tourniquet. This is the first application of the tourniquet.
   * Upon the completion of the tourniquet application, the blinded observer records the presence or absence of a dopplerable pulse. A blinded observer again uses a doppler ultrasound probe to check the dorsalis pedis (DP) pulse, the artery pulse on the surface of the foot, at the previously marked "X" location on the foot.
   * The medical professional removes the tourniquet and the study participant takes a break.
   * The medical professional places a blood pressure cuff first and then places a tourniquet over the blood pressure cuff. This is the second application of the tourniquet. The blood pressure cuff will be attached to a pressure sensor to measure surface pressure under the tourniquet. The medical professional will tighten the tourniquet until the doppler pulse is eliminated. The medical professional will then read and record the pressure readings.
   * The medical professional removes the tourniquet.

   The procedures will then be repeated to a participant's other leg for the other arm. For example, if a participant is initially assigned to the CAT and uses the right leg for tourniquet application. The participant will then be in the LAVA TQ arm for the left leg.

   Termination Procedures: For the first tourniquet application on each leg, the observer will use doppler ultrasound to assess the participant's foot for a present or absent dorsalis pedis pulse. The observer will make the assessment at the location previously marked with a surgical marker. As soon as the pulse is determined to be present or absent, the observer will verbally tell the medical professional, "remove the tourniquet now."

   For the second tourniquet application on each leg, the medical professional will tighten the tourniquet on top of the neonatal blood pressure cuff as described. The study team member will record the pressure. As soon as the pressure is noted, the study team member will tell the medical professional, "remove the tourniquet now."

   Participant Post-Application Assessment: Following the application of two tourniquets to both legs, the study team will ask the participant to rest while lying on the table for five minutes. After five minutes, the study team member will ask the participant the following questions:
   * Do you have any persistent pain beyond mild aching at the application site?
   * Do you have numbness, tingling, or other abnormal sensations?
   * Does your leg feel weak?

   If the answer is yes to any question, the team member will ask the participant to rest for five more minutes and re-ask the questions. If the answer to any question is still yes, the study team member will recommend that the participant seek medical care at an emergency department or with the participant's physician. If the study team member or participant is concerned that they are experiencing a medical emergency, they will call 9-1-1 and alert any of the medical professionals assisting with the study for assistance.

   If the answer to the questions is no, the study team member will ask the participant to walk up and down the hall in the MDL. The study team member will observe the participant ambulating. If the person feels normal while walking, they can be discharged from the study.

   The study team member will be advised to follow-up with their physician or emergency department for medical care if either leg develops worsening pain, swelling, redness, coldness, or bluish or pale color, or if they have shortness of breath or chest pain. The study team member will advise the participant that some mild local bruising or redness in the area of the tourniquet application may occur and that it does not require medical evaluation.

   In addition, given the LAVA TQ is an abbreviated investigational device, we will follow the abbreviation requirements specified by the FDA.
4. Data Collection

   The outcome variables in the study are: 1. the participants' resting blood pressure, 2.

   the presence or absence of dorsalis pedis pulse after tourniquet application, and 3. the surface pressure reading when the tourniquet is tightened. At the beginning of the study, participants will be asked to complete a demographic information sheet. On this sheet, they will fill out their age, gender, race, and ethnicity.
5. Statistical Considerations

The primary outcome variable for this research study binary (successfully stop the pulse: yes/no) and we conducted a power analysis for a parallel group non-inferiority trial. Assuming the two arms have the same high successful rate, with 80% power, and define the non-inferiority limit as 10% (so that a difference bigger than this would matter in practice), we estimated sample size required for each group is 13 applications (at least), so a total sample size of 26 applications (at least). Given the potential missing data and to ensure we will have enough statistical power for the final analyses, we will set the total sample size of 40 applications for this study. Since the tourniquet will be applied to participants' both legs (not at the same time), each leg will be one application and one participant will be able to fulfill two applications. As such, we will recruit no more than 20 participants for the study session and one additional participant for the training session.

ELIGIBILITY:
Inclusion Criteria:

* The study population includes individuals with access to the USU campus and prior tourniquet experience (an individual has received tourniquet training previously or has used tourniquet before so that they would understand the discomfort when a tourniquet is applied).

Exclusion Criteria:

* Individuals with the following conditions or history will be excluded from participation: hypertension, prior vascular surgery, peripheral vascular disease, diabetes, prior lower extremity vascular surgery, active lower extremity infection, any hypercoagulable condition (such as Factor V Leiden, or Protein C and S deficiency), pregnancy, or any condition in which the participant is concerned they may suffer harm from brief tourniquet application.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Successful occlusion | While tourniquet is applied to leg (application 1)
  Successful occlusion of blood flow is indicated by the absence of the dorsalis pedis pulse, as measured by a Doppler ultrasound.

SECONDARY OUTCOMES:
Applied pressure | While tourniquet is applied to leg (application 2)
  Surface pressure under the tourniquet when applied, as measured by a neonatal blood pressure cuff attached to a pressure sensor system

CONTACTS AND LOCATIONS:
Overall Officials: Craig Goolsby, MD, MEd, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Uniformed Services University of the Health Sciences, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Levy MJ, Jacobs LM. A Call to Action to Develop Programs for Bystanders to Control Severe Bleeding. JAMA Surg. 2016 Dec 1;151(12):1103-1104. doi: 10.1001/jamasurg.2016.2789. No abstract available. PMID 27626623
- [Background] Lei R, Swartz MD, Harvin JA, Cotton BA, Holcomb JB, Wade CE, Adams SD. Stop the Bleed Training empowers learners to act to prevent unnecessary hemorrhagic death. Am J Surg. 2019 Feb;217(2):368-372. doi: 10.1016/j.amjsurg.2018.09.025. Epub 2018 Sep 26. PMID 30292328
- [Background] Kragh JF Jr, O'Neill ML, Walters TJ, Jones JA, Baer DG, Gershman LK, Wade CE, Holcomb JB. Minor morbidity with emergency tourniquet use to stop bleeding in severe limb trauma: research, history, and reconciling advocates and abolitionists. Mil Med. 2011 Jul;176(7):817-23. doi: 10.7205/milmed-d-10-00417. PMID 22128725

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/33/NCT05504733/Prot_SAP_ICF_000.pdf